CLINICAL TRIAL: NCT01327963
Title: Long-term Outcomes After Transoral Incisionless Fundoplication (TIF) Performed in Routine Clinical Practice: The Retro TIF Study
Brief Title: Retrospective TIF Study for Treatment of Gastroesophageal Reflux Disease (GERD). The RetroTIF Study
Acronym: RetroTIF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor is focusing on prospective randomized studies
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D01079
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal reflux disease; GERD; Heartburn; Reflux; Regurgitation; Hoarseness; Cough
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Hoarseness; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transoral Incisionless Fundoplication (Experimental): Intervention: Transoral Incisionless Fundoplication 2.0 technique iteration (TIF 2.0).
  With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro-esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GastroEsophageal Junction (GEJ) below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Interventions: Device: Transoral Incisionless Fundoplication

INTERVENTIONS:
Device: Transoral Incisionless Fundoplication — Transoral incisionless esophago-gastric fundoplication performed using the EsophyX (brand name) system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized Transoral Incisionless Fundoplication 2.0 technique iteration (TIF2.0) protocol.
  Other Names: TIF

SUMMARY:
The purpose of this retrospective, open-label, post-market study is to evaluate the safety and efficacy of Transoral Incisionless Fundoplication (TIF) performed with EsophyX (brand name) in a broad range of GastroEsophageal Reflux Disease (GERD) patients treated at high volume centers across the United States.

DETAILED DESCRIPTION:
This retrospective, open-label, post-market study evaluates the safety and efficacy of Transoral Incisionless Fundoplication (TIF) performed with EsophyX (brand name) in a broad range of GastroEsophageal Reflux Disease (GERD) patients treated at high volume centers across the United States, in clinical routine practice, as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* Have undergone the TIF procedure within the past 2 years
* History of daily proton pump inhibitor (PPI) use for >6 months
* Proven gastroesophageal reflux by either endoscopy, ambulatory potential of hydrogen (pH) or moderate to severe symptoms on or off PPIs
* Deteriorated gastroesophageal junction (Hill grade II or III)
* Availability for a follow-up visit at 6,12 or 24 months
* Willingly and cognitively signed informed consent

Exclusion Criteria:

* Procedure not completed or performed following a non-standardized TIF protocol
* Subjects suffering from other gastrointestinal (GI) conditions such as dyspepsia, celiac disease, Irritable bowel syndrome (IBS) or Crohn's disease
* Pregnancy
* Enrollment in another device or drug study that may confound the results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Barnes, MD MBA FACS, Principal Investigator — Livingston Hospital and Healthcare Services Inc, CAH
Locations (2):
- United States (2):
  - Munroe Regional Medical Center, Ocala, Florida
  - Livingston Hospital and Healthcare Services, Inc. CAH, Salem, Kentucky

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 124 patients were eligible to participate in the study, but 110 signed consent and started the study. Of the 14 that didn't start, 13 could not be reached at start of study and one patient did not receive the TIF procedure due to intraoperative hematoma.
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication 2.0 technique iteration (TIF 2.0).
  With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro-esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the Gastroesophageal Junction (GEJ) below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX (brand name) system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized transoral incisionless fundoplication 2.0 technique iteration (TIF2.0) protocol.
Period: Overall Study
Arm/Group | Transoral Incisionless Fundoplication
Started | 110
Completed | 110 (110 participants signed informed consent to be included in the study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is 110 of 124 who were eligible. 110 signed informed consent to participate in the study.
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication: TIF 2.0 technique iteration.
  With patient in general anesthesia. The EsophyX device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro -esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GEJ below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX (brand name) system with SerosaFuse (brand name) prolene fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized TIF2.0 protocol.
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 110
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 29
Region of Enrollment [Number; unit: participants] — 64 patients from Livingston Hospital and Healthcare Services in Salem, Kentucky, and 60 from Munroe Regional Medical Center in Ocala, Florida were eligible to participate in the study but 110 signed consent and started. 13 eligible patients were lost to follow up at start of study, and one did not have Transoral Incisionless Fundoplication (TIF) completed due to intraoperative hematoma.
  participants
    United States | 110
Body Mass Index (BMI) > or equal to 35 [Count of Participants; unit: Participants] | 18
Gastroesophageal Reflux disease (GERD) symptom duration (years) [Count of Participants; unit: Participants] — median number of years of GERD symptom duration is 9 years
  Participants
    1-2 years | 13
    2-5 years | 14
    > or equal to 5 years | 83
Proton Pump Inhibitor (PPI) therapy duration (years) [Count of Participants; unit: Participants] — median number of years of PPI duration therapy is 8 years
  Participants
    1-2 years | 16
    2-5 years | 13
    > or equal to 5 years | 81
Hiatal hernia size [Count of Participants; unit: Participants] — This is a subjective measure made by the study investigator using endoscopic visualization of the gastroesophageal junction. Normal or small hiatal hernia is <= 1cm. Hill Grade system is used: Hill I, II, III, IV, with Hill I normal hiatus and Hill IV large, loose hiatal opening. Hill IV is an exclusion for this study.
  Hill II may indicate a 2cm hiatal hernia, Hill III a 3cm hiatal hernia for example. Population: 70 of 110 participants had a 2 or 3cm hiatal hernia at baseline
  Participants
    number analyzed (Participants) | 70
    2cm hiatal hernia (sliding) | 51
    3cm hiatal hernia (sliding) | 19
Esophagitis using Los Angeles (LA) grading [Count of Participants; unit: Participants] — LA grading of esophagitis is an A, B, C, D system, where A is the least severe esophagitis and D is the most severe. LA grade D is an exclusion for this protocol. Normal or no esophagitis reported, will have no grade listed. LA grading is a subjective measure made using an endoscope to visualize the gastroesophageal junction to assess for esophagitis based on the LA grade criteria. An improvement of one grade post-TIF is considered a success, e.g., from grade B to grade A, or grade A to no grade (normal), etc. Population: 64 of 110 participants had esophagitis at baseline
  Participants
    number analyzed (Participants) | 64
    LA grade A | 42
    LA grade B | 20
    LA grade C | 2

OUTCOME MEASURES:

1. Primary Outcome: Typical and Atypical Gastroesophageal Reflux Disease (GERD) Symptom Elimination
Description: Typical and atypical GERD symptom elimination in GERD Health-Related Quality of Life (GERD-HRQL). HRQL questionnaire measures typical GERD symptoms, scale 0-5 for each of 9 questions; scores considered normalized if every score is 0), GERD Symptom Score (GERSS measures atypical GERD symptoms, scale 0-3 for severity and 0-4 for frequency, with total scale 0-60; patients with controlled reflux symptoms are expected to have a score of <18) and Reflux Symptom Index (RSI measures atypical laryngopharyngeal (LPR) symptoms, scale 0-5 for each of 9 questions with maximum of 45 with a normality threshold of < or = 13) questionnaires) at the follow-up.
Time Frame: median 7 months (range 5-17 months)
Measure: Count of Participants; unit: Participants
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication: TIF 2.0 technique iteration.
  With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro -esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GEJ below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized Transoral Incisionless fundoplication 2.0 technique iteration (TIF2.0) protocol.
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 110
Participants
  Participants with normal GERD-HRQL scores | 88
  Participants with controlled reflux symptoms measured by GERSS questionnaire | 87
  Patients scoring in the normality threshold on RSI questionnaire | 83

2. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs) & Unanticipated Adverse Device Effects (UADEs)
Description: The treatment will be considered safe if the incidence of serious adverse events (SAEs) is below the ranges reported for laparoscopic fundoplication.
Time Frame: median 7 months (range 5-17 months)
Population: There were no serious adverse events or UADE during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication 2.0 iteration (TIF 2.0). With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro -esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GEJ below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized TIF2.0 protocol.
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 110
Participants | 0

3. Secondary Outcome: Number of Participants Reporting Complete Elimination of Proton Pump Inhibitor (PPI) Use
Description: Patients reporting complete discontinuation of daily PPI use will be considered clinically significant.
Time Frame: median 7 months (range 5-17 months)
Measure: Count of Participants; unit: Participants
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication 2.0 technique iteration (TIF 2.0).
  With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro -esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GEJ below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX (brand name) system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized TIF2.0 protocol.
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 110
Participants | 102

4. Secondary Outcome: Number of Participants With Healing of Reflux Esophagitis
Description: One LA grade reduction will be considered clinically significant. LA grades are A, B, C, D, with A being the least severe esophagitis. No grade assigned is considered "normal", i.e. no esophagitis reported.
Time Frame: median 7 months (range 5-17 months)
Population: Of 53 patients examined at follow up for esophagitis or hiatal hernia status, 30 had reported esophagitis at baseline. Please note: there was 1 new case of esophagitis reported at follow-up, that had not been present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 30
Participants | 25

5. Secondary Outcome: Number of Participants Whose Baseline Hiatal Hernia Has Remained Reduced at Post-TIF Follow-up
Description: Measurement obtained by study investigator, under endoscopic visualization using cm markings on the endoscope. Outcome measure assesses if hiatal hernia that was present at baseline and reduced (size reduction to < 1 cm is considered clinically significant) during TIF procedure, has remained reduced at the post-TIF follow up exam.
Time Frame: median 7 months (range 5-17 months)
Population: 53 patients were assessed for esophagitis and presence of hiatal hernia at follow-up. Hiatal hernia was present at baseline and reduced during TIF procedure in 34 of the patients examined at follow-up. Hiatal hernia in 33 of 34 remained reduced at follow-up. Please note: there was one new case of hiatal hernia reported that had not been present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 34
Participants | 33

6. Secondary Outcome: Number of Participants With Normalization or Clinically Significant Improvement in Esophageal Acid Exposure Assessed by Impedance/pH Testing and Reflux Episodes
Description: Esophageal acid exposure will be measured objectively by 48-hour Bravo Potential of Hydrogen (pH) or 24-hour impedance/pH testing at the follow-up (where pH testing is available). Normalization of esophageal acid exposure will be defined by total time pH< 4 for ≤ 6% of 24-hour or for ≤ 5.3% of 48-hour monitoring period. The number of reflux episodes of ≤ 44 per each 24-hour period will be considered normal.
Time Frame: median 7 months (range 5-17 months)
Population: Note: neither 48-hour Bravo pH nor 24-hour impedance/pH testing was completed. pH testing was unavailable at the study sites. Study protocol noted that testing would be completed "if available". In the absence of these testing tools, sites relied on detailed history, physical signs, symptom evaluation, barium swallow, and repeated esophagogastroduodenoscopy (EGD) with biopsy to make diagnosis. This continues to be the most commonly used method of GERD diagnosis among community physicians.
Arm/Group | Transoral Incisionless Fundoplication
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: This is a retrospective study. TIF procedures were performed from November 2008 through December 2009. The study enrolled patients and collected post-TIF follow up visits in 2010. Adverse event data was collected from day of TIF procedure through final follow-up visit.
Description: There was an intra-op event described in the study publication, but because the TIF procedure could not be completed due to an intra-op hematoma, patient did not sign consent or start this retrospective study. This is not included as a study-related adverse event.
Groups:
- Transoral Incisionless Fundoplication: Intervention: Transoral Incisionless Fundoplication 2.0 technique iteration (TIF 2.0).
  With patient in general anesthesia. The EsophyX (brand name) device is introduced through the mouth, over a standard endoscope, into the stomach. Multiple gastro-esophageal plications are performed, apposing the fundus to the distal part of the esophagus and repositioning the GEJ below the diaphragm, into the abdomen. Multiple prolene fasteners are used to secure and keep in place the plications.
  Transoral Incisionless Fundoplication: Transoral incisionless esophago-gastric fundoplication performed using the EsophyX (brand name) system with SerosaFuse (brand name) fasteners (EndoGastric Solutions, Inc., Redmond, Washington, USA) and following the standardized TIF2.0 protocol.
Arm/Group | Transoral Incisionless Fundoplication
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No